CLINICAL TRIAL: NCT02506569
Title: ProMRI 3T ENHANCED Master Study
Status: Completed | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: TA109
Record Dates: First submitted 2015-07-14; First posted 2015-07-23 (Estimated); Last update posted 2018-02-07 (Actual); Status verified 2018-02

CONDITIONS: Safety of MR (Magnetic Resonance)-Conditional ICDs
MeSH Terms: interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Implantable Cardioverter Defibrillator therapy — Tachycardia Fast Heart Beat
Other: Magnetic Resonance Imaging (MRI) — MRI scan of the head and lower body parts

SUMMARY:
The investigation is designed to provide supporting evidence for the clinical safety of the Biotronik's new Implantable Cardioverter Defibrillator systems when used under specific 3 Tesla MR conditions .

ELIGIBILITY:
Inclusion Criteria:

* Implanted with Implantable Cardioverter Defibrillator (ICD) system according to Clinical Investigational Plan (CIP)
* ICD system was implanted in the pectoral region
* Implantation at least 5 weeks prior to enrollment date
* Patient body height ≥ 140 cm
* Age ≥ 18 years
* Right Ventricular pacing threshold (at 0.4 ms) measurable and ≤ 2.0 V
* Written informed consent
* Able and willing to complete MRI testing
* Able and willing to complete all testing required by the clinical protocol
* Available for all follow-up visits at the investigational site

Exclusion Criteria:

* Standard contraindication for MRI scans
* Patient shows signs of a twiddler's syndrome, i.e. fiddles with implant
* Explantation, exchange or reposition of ICD or lead within 5 weeks prior to enrollment date
* Charging status of the battery is Elective Replacement Indicator (ERI) or End of Service (EOS)
* MRI scan within 5 weeks prior to enrollment date
* R-wave sensing amplitude < 6.5 millivolt
* Lead impedance less than 200 or greater than 1500 Ohm
* Life expectancy of less than six months
* Cardiac surgery in the next six months
* Pregnant or breastfeeding
* Participation in another interventional clinical investigation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients selected for participation should be from the investigator's general patient population according to the inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2015-01; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Serious Adverse Device Effect (SADE)-free rate of implantable cardioverter defibrillators and leads possibly or securely related to the MRI procedure | 1 Month
Increase in pacing thresholds ratios measured between 1-month post-MRI and pre-MRI | 1 Month
  Evaluate the percentage of ICD leads with an increase in the pacing threshold ratio measured between the Pre-MRI and 1-month post-MRI
Decrease in sensing amplitude ratios between 1-month post-MRI and pre-MRI | 1 Month
  Evaluate the percentage of ICD leads with a decrease in the sensing amplitude ratio measured between the Pre-MRI and 1-month post-MRI

CONTACTS AND LOCATIONS:
Overall Officials: Rainer Zbinden, Dr., Principal Investigator — Triemli Hospital
Locations (12):
- Australia (3):
  - Flinders Medical Centre, Bedford Park
  - Royal North Shore Hospital, Sydney
  - Westmead Hospital, Westmead
- Austria (2):
  - Allgemeines Krankenhaus Linz, Linz
  - Landesklinikum St. Pölten, Sankt Pölten
- Germany (5):
  - Deutsches Herzzentrum Berlin, Berlin
  - Klinikum Coburg, Coburg
  - Uniklinikum Düsseldorf, Düsseldorf
  - Universitätsklinikum Göttingen, Göttingen
  - St. Bonifatius Hospital, Lingen
- National Heart Centre, Singapore, Singapore
- Stadtspital Triemli, Zurich, Switzerland